CLINICAL TRIAL: NCT05925335
Title: Evaluation of Clinical Outcomes of Transseptal Transcatheter Mitral Valve-in-Valve Replacement for Degenerated Bioprostheses - The China Mviv Registry
Brief Title: The China Mviv Registry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Yan Wang, Xiamen Cardiovascular Hospital, Xiamen University, Xiamen Cardiovascular Hospital, Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YLK 21
Record Dates: First submitted 2023-05-11; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Bioprosthesis Failure; Mitral Stenosis With Insufficiency; Mitral Stenosis; Mitral Regurgitation; Heart Failure
MeSH Terms: conditions — Mitral Valve Stenosis; Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcatheter mitral valve-in-valve implantation (Experimental)
  Interventions: Device: Transseptal Transcatheter Mitral valve-in-valve Replacement

INTERVENTIONS:
Device: Transseptal Transcatheter Mitral valve-in-valve Replacement — Transcatheter transfemoral mitral valve-in-valve replacement is an alternative surgery in patients with severe dysfunction of a degenerated mitral bioprosthesis and high surgical risk for repeat operation. The procedure is performed via femoral vein access. All procedures were carried out using intra-procedural TEE guidance to aid in transseptal puncture. After balloon septostomy, the bioprosthetic valve is introduced through the degenerative valve into the left ventricle and expanded in the mitral position during rapid ventricle pacing.

SUMMARY:
Mitral valve disease is the most common structure heart disease, and surgical valve replacement is an important treatment for severe mitral valve disease. There are 2 types of valve often been used, mechanical or biological protheses valves. Mechanical valve requires lifelong use of anticoagulants and take the risk of bleeding through all lifetime, but bioprotheses valve do not..

DETAILED DESCRIPTION:
Due to a massive shift from mechanical to bioprosthetic valves with finite longevity, increasing numbers of patients are presenting with bioprosthetic mitral valve degeneration. Mitral valve reoperation, the standard therapy for the bioprosthetic failure in the past, often entails high risk due to age, multiple comorbidities et al. TMVR is an emerging treatment for the patients with bioprosthetic failure at high risk for conventional mitral valve surgery. Recent studies from US and Europe have demonstrated the safety and efficacy of TMVR in this population. However, there are limited data regarding clinical outcomes after TMVR from Asia-Pacific region. To evaluate the safety and efficacy of TMVR using balloon-expandable valve among those patients with high risk for redo surgery and those who refuse redo surgery after shared decision making even they have less than high risk.

ELIGIBILITY:
Inclusion Criteria:

* Subject had a degenerated surgical mitral bioprosthesis with at least moderate to severe mitral regurgitation or severe stenosis with echocardiographically derived mitral valve area (MVA) of ≤1.5 cm2
* Subjiect is symptomatic from mitral valve disease, as demonstrated by reported NYHA Functional Class II or greater.
* Subject is at least 18 years old.
* Heart team (including cardiac surgeon) agree on eligibility including assessment that transeptal, transcatheter mitral valve replacement (TsMVR) and redo surgical mitral valve replacement (rSMVR) are appropriate.
* The study patient or the study patient's legal representative informed of the nature of the study, agreed to its provisions and provided written informed consent as approved by the Institutional Review Board (IRB) center.
* The study Subject agreed to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which was conducted as a phone/clinic follow-up.

Exclusion Criteria:

* Subject was operable with the assessment of experienced Heart Team
* Subject had evidence of an acute MI, percutaneous intervention, or a peripheral intervention ≤30 days prior to Portico ViV index procedure.
* Subject had uncontrolled blood dyscrasias defined as: leukopenia (WBC<3,000 mm3), acute anemia (Hb <9 g/dL), or thrombocytopenia (platelet count <50,000 cells/mm³).
* Subject was considered hemodynamically unstable at the time of the ViV procedure (requiring inotropic support or mechanical heart assistance)
* Subject had severe ventricular dysfunction with left ventricular ejection fraction (LVEF) <20% as measured by resting echocardiogram.
* Subject had imaging evidence of intracardiac mass, thrombus or vegetation.
* Subject had an active peptic ulcer or has/had upper gastrointestinal (GI) bleeding ≤3 months prior to ViV index procedure.
* Subject had a documented history of a cerebrovascular accident (CVA) or a transient ischemic attack (TIA) ≤6 months prior to index procedure.
* Subject had active bacterial endocarditis or ongoing sepsis ≤ 6 months prior to the index procedure.
* Subject was unable to tolerate antiplatelet or anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-11 (Estimated); Primary Completion 2024-07-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 12 months
  The rate in all-cause mortality will be calculated from 0 month to 12 months.
Rate of New hospitalization for heart failure | 12 months
  Hospitalization for valve-related symptoms or worsening congestive heart failure

SECONDARY OUTCOMES:
Technical success | 24 hours
  Technical success was the primary safety endpoint at the time of patient exit from the cardiac catheterization laboratory, which was defined as the delivery and retrieval of the transcatheter delivery system being successful, the deployment of a single valve in the proper position in the mitral annulus, no need for surgery or additional reintervention, and the patient leaving the procedure room alive
Procedure success | 12 months
  Procedure success defiened as adequate performance of the THV with residual MR grade < 2 and mean MV gradient (MVG) < 10 mm Hg.
all-cause mortality | annual for five years
  The rate in all-cause mortality will be calculated from 0 month to 12 months.
Rate of New hospitalization for heart failure | annual for five years
  Hospitalization for valve-related symptoms or worsening congestive heart failure
Rate of myocardial infarction | annual for five years
Rate of neurological events | annual for five years
  All stroke, transient ischemic attack (TIA)
Rate of Structural Valve dysfunction | annual for five years
  as assessed by transthoracic echocardiography with residual MR grade > 2 and mean MV gradient (MVG) ≥ 10 mm Hg.
Clinical Benefit Endpoint | 30 days, 6 months, 12 months, annual for five years]
  Change in New York Heart Association (NYHA) functional classification from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Dr, Principal Investigator — Clinical Trial Center of Xiamen Cardiovascular Hospital
Locations (1):
- Yan Wang, Xiamen, Fujian, China